CLINICAL TRIAL: NCT01853007
Title: Communicating About Choices in Transplantation (COACH)
Brief Title: Communicating About Choices in Transplantation
Acronym: COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PD301152
Record Dates: First submitted 2013-05-07; First posted 2013-05-14 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: End Stage Renal Disease and Kidney Transplantation
Keywords: End stage renal disease; Kidney transplantation; Transplant options (living and deceased donor); Patient education; Communication skills training
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients in this arm will receive only the education offered by the transplant center, as required by Medicaid. Upon completion of all data collection activities, patients in this arm will be offered the program.
- COACH Program (Experimental): Participants randomized to the intervention condition will attend a COACH session held in a small group format. The session provides information on living and deceased donor transplantation (i.e., the processes, risks and benefits) and on the key communication skills needed to effectively initiate and maintain conversations about transplantation.
  Interventions: Behavioral: COACH Program

INTERVENTIONS:
Behavioral: COACH Program
  Arms: COACH Program

SUMMARY:
The purpose of this study is to test the impact of a newly developed educational program on kidney transplant candidates' communication about living and deceased donor kidney transplantation.

DETAILED DESCRIPTION:
The Communicating about Choices (COACH) in Transplantation program educates patients with end stage renal disease, who are waitlisted for kidney transplantation, about kidney disease and the risks, benefits and processes for both living and deceased donor transplantation. The program also teaches key communication skills needed to effectively initiate and manage conversations about transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Wait listed for kidney transplantation in active status
* Adult (at least 18 years of age)
* English speaking
* Capable of making medical decisions (i.e., not cognitively impaired)
* Non-institutionalized

Exclusion Criteria:

* Not listed for kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in engagement in discussion of living and deceased donor transplantation | Baseline (upon enrollment); 1 month post; 3 months post
  2 self-report items: whether transplantation was discussed (yes/no) and the number of discussions held
Change in knowledge of living and deceased donor transplant | Upon enrollment (baseline); 1 month post; 2 months post
  15 True/False Questions

SECONDARY OUTCOMES:
Change in intentions to discuss living and deceased donor transplantation | Upon enrollment (baseline); 1 month post; 3 months post
  3-item, 7-point Likert-type scale

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Traino, PhD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States